CLINICAL TRIAL: NCT06073041
Title: Implementing and Evaluating the Comprehensive Integration of Physical Activity Into a Major Health System and Connecting Patients to Community-based Physical Activity Programs
Brief Title: Implementing and Evaluating the Integration of Physical Activity Into a Major Health System and Connecting Patients to Physical Activity Programs.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Temple University (Other); University of Utah (Other); University of Nebraska (Other); Durham University (Other)
Responsible Party: Principal Investigator, Jennifer Trilk, Professor, University of South Carolina
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R56HL157218-01A1 (NIH)
Record Dates: First submitted 2023-09-18; First posted 2023-10-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chronic Disease; Exercise; Physical Activity
Keywords: Physical activity; Evidence-based; Exercise; RE-AIM; Implementation; Adoption; Referral pathway
MeSH Terms: conditions — Chronic Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: All eligible clinics were invited to adopt the EIMG model (primary aim). Those that adopted the EIMG model received a sequential intervention involving onboarding and implementation (secondary aim).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adopter (Experimental): Clinics that decide to adopt the EIMG Program
  Interventions: Other: Invitation to adopt; Behavioral: Onboarding strategies
- Non Adopter (Other): Clinics that decide not to adopt the EIMG Program
  Interventions: Other: Invitation to adopt

INTERVENTIONS:
Other: Invitation to adopt — All eligible Prisma Health clinics will be invited to adopt EIMG.
Behavioral: Onboarding strategies — Providers at adopting clinics will first be sent an instructional video as a part of a low touch initial onboarding (phase 1). After 4 months, clinics will then receive an in-depth standardized onboard training (phase 2).
  Arms: Adopter

SUMMARY:
Multiple case study trial examining the adoption, implementation, and reach of eligible patients visiting participating Prisma Health primary care clinics and receiving a referral to a 12-week evidence-informed physical activity (PA) program hosted at local community PA facilities.

DETAILED DESCRIPTION:
This study will employ a single arm, multiple case study design using a mixed methods approach to examine the adoption, implementation, and reach of EIMG across Prisma Health primary care clinics (i.e., clinic workflow, referral process), leading to patient enrollment in a community-based, evidence-informed PA program. Eligible Prisma Health primary care clinics that have not yet received EIMG onboard training and activation will be provided with the opportunity to adopt EIMG as a part of their clinic practice and patient workflow process. A mixed methods approach will examine contextual factors influencing decisions to adopt/not adopt EIMG.

Clinic champions at clinics adopting EIMG will be provided with a brief pre-recorded training video to disseminate to their clinic staff on how to provide their patients with an EIMG referral (phase 1). All providers at the clinic will have the ability to screen and identify physically inactive patients and provide them with an EIMG referral. Initial implementation and reach of EIMG at adopting clinics will be tracked for approximately four months following the dissemination of the pre-recorded training video. After four months, the EIMG team will provide a more in-depth, standardized clinic onboard training following established protocols iteratively developed and refined through the initial addition of EIMG clinics between 2016-19 (phase 2). The onboard training, which consists of an overall presentation of the EIMG program and specific information on placing the referral order and patient workflow, has been adapted for virtual environments due to its notable added benefits, including its recording to serve as an ongoing reference tool for those who cannot attend initial training and incoming staff. Implementation and reach of EIMG will be tracked for an additional four months after the onboard training.

Referred patients will have the opportunity to enroll in an evidence-informed, 12-week PA program at local community PA facilities (e.g., YMCAs) that partner with EIMG. Upon enrollment and at the completion of the 12-week PA program, patients will undergo an assessment battery that includes the completion of a patient health questionnaire, anthropometric assessments (i.e., height, weight, waist circumference) and an evaluation of their mental and emotional health (i.e., PROMIS tool, PHQ-9). The RE-AIM framework will inform the assessment of implementation outcomes (i.e., adoption, implementation, and reach), while the i-PARIHS framework will be used to examine contextual factors (i.e., determinants) influencing clinic level outcomes. Patient demographics, health outcomes, healthcare utilization and costs of eligible patients at participating primary care clinics, both before and after EIMG onboarding, will be extracted from the Prisma Health electronic health record (EHR) system. Data will be compared between patients that receive EIMG referrals and matched controls at clinics that do not adopt EIMG: 1) the impact of EIMG on changes in health outcomes, and 2) the impact of EIMG on healthcare costs. These estimates will be used as the basis for cost-effectiveness analyses of EIMG and serve as the foundation for long-term evaluation modeling approaches to incorporate changes in longer-term secondary health outcomes (e.g., stroke, acute myocardial infarction) on healthcare costs.

ELIGIBILITY:
Clinic Inclusion Criteria:

* Prisma Health primary care clinic (i.e., family or internal medicine) located in the Upstate of South Carolina
* At least two attending providers

Clinic Exclusion Criteria:

* Clinics greater than 15 miles from a participating community physical activity facility
* Have received EIMG onboarding or activation in the past

Clinical Staff Inclusion Criteria:

* Prisma Health employed
* Actively seeing patients at an activated EIMG clinic by the beginning of the phase in which they will be enrolled in the study (providers)
* Staff member at an activated EIMG clinic by the beginning of the phase in which they will be enrolled in the study (managers/clinic staff)

Clinical Staff Exclusion Criteria:

* Less than 18 years old

Patient Inclusion Criteria:

* Have received an EIMG referral from their primary care provider beginning September 5, 2023

Patient Exclusion Criteria:

* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Adoption of EIMG at eligible primary care clinics | Months 0-1
  Rate of EIMG adoption at eligible primary care clinics

SECONDARY OUTCOMES:
Factors in decision to adopt/not adopt EIMG | Months 1-2
  Interviews with clinic managers at adopting and non-adopting clinics
Referral of eligible patients to EIMG in adopting clinics (phase 1) | Months 1-4
  Number of referrals given to EIMG-eligible patients by providers in adopting clinics
Referral of eligible patients to EIMG in adopting clinics (phase 2) | Months 5-8
  Number of referrals given to EIMG-eligible patients by providers in adopting clinics
Feedback on EIMG referrals and onboarding strategies from clinic staff | Months 9-12
  Interviews with clinic staff members at adopting clinics
Patient physical activity levels (minutes of moderate-to-vigorous activity/week) | Conducted at months 0, 1.5, 3, 9, 15
  Assessing changes in patient physical activity levels via the Physical Activity Vital Sign. Assessments will occur prior to enrollment in the 12-week physical activity program (week 0), midway through the program (week 6), at the completion of the program (week 12), as well as long-term maintenance (conducted via phone call 6- and 12-months post-program)
Patient blood pressure levels (mmHg) | Months 1-16
  Assessing changes in patient blood pressure using a digital blood pressure monitor. Assessments will occur prior to enrollment in the 12-week physical activity program (week 0), midway through the program (week 6), at the completion of the program (week 12). Additional blood pressure measurements may also be extracted from the Prisma Health electronic health records for the time period six months before and twelve months after the 12-week physical activity program.
Patient bodyweight (kg) | Months 1-16
  Assessing changes in patient bodyweight using a minimum of a class III category weighing scale. Assessments will occur prior to enrollment in the 12-week physical activity program (week 0), midway through the program (week 6), and at the completion of the program (week 12). Additional bodyweight measurements may also be extracted from the Prisma Health electronic health records for the time period six months before and twelve months after the 12-week physical activity program.
Impact of EIMG on healthcare costs | Months 1-16
  Using data from the Prisma Epic electronic health record (EHR), we will extract primary health outcomes (e.g., blood pressure, body weight, hemoglobin A1c, lipid profiles) from the index (first) visit and again at the end of a care episode for all patients who received an EIMG referral at participating clinics during the study period. We will use the EHR record to assess changes in outcomes across the care episode and all healthcare utilization for each patient during the care episode to estimate costs. This approach will yield estimates of: 1) the impact of EIMG on changes in health outcomes across the care episode, and 2) the impact of EIMG healthcare costs during the care episode. We will use these estimates for a short-term cost-effectiveness analysis of the EIMG program, as well as the foundation for long term evaluation for modeling approaches changes in longer-term secondary health outcomes (e.g., stroke, acute myocardial infarction) on healthcare costs.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Trilk, PhD, Principal Investigator — University of South Carolina; Mark Stoutenberg, PhD, Principal Investigator — Durham University
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Scientific data that will be preserved and shared: individual interviews, online surveys, electronic health record data.
  The raw data collected for the individual interviews, online surveys, and clinical data will be electronically stored in a secured, cloud-based storage. Identifiers will be removed and maintained in a separate secure file for future reference. Patient information extracted from the Prisma Health EHR will be de-identified by the honest broker/data analyst before secure transfer to the research team. Sharing of this data will follow guidelines established by the Prisma Health Office of Research and Innovation.
Supporting Information: Study Protocol, SAP
Time Frame: All data will be made available at the completion of the project, no later than the time of publication. The duration of preservation and sharing of the data will be in perpetuity.
Access Criteria: All data (online survey data, interview data, program participant data, and EHR data) will be de-identified and stored in data sharing repository, such as the Open Science Framework (OSF) or the Biologic Specimen and Data Repository Information Coordinating Center (BIOLINCC) managed by NHLBI.
  We will use unique persistent identifiers to improve data findability. The data sharing repository will provide metadata and assign our dataset a digital object identifier for ease of access.

REFERENCES:
- [Derived] Stoutenberg M, Estabrooks PA, Brooks JM, Jindal M, Wichman C, Rosemeyer J, Schumacher LM, McNulty LK, Ewing A, Eskuri S, Bennett F, Trilk JL. Implementing and evaluating the comprehensive integration of physical activity into a major health system: study design and protocol. BMJ Open. 2025 Jan 6;15(1):e091556. doi: 10.1136/bmjopen-2024-091556. PMID 39762113

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT06073041/Prot_SAP_000.pdf